CLINICAL TRIAL: NCT00001343
Title: The Relative Effects of Androgen, Estrogen, and the Combination of Androgen and Estrogen on Growth Rate, GH Binding Protein, IGF-I, and Cognitive Function in Growth Hormone-Treated Girls With Turner Syndrome
Brief Title: The Effects of Hormones in Growth Hormone-Treated Girls With Turner Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930054; 93-CH-0054
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-10

CONDITIONS: Dwarfism; Turner's Syndrome
Keywords: Turner's Syndrome; Short Stature; Cognitive Function; Sex Steroids; Turner Syndrome; TS
MeSH Terms: conditions — Dwarfism; Turner Syndrome | interventions — Human Growth Hormone; Oxandrolone

INTERVENTIONS:
Drug: Humatrope
Drug: Oxandrolone

SUMMARY:
Turners Syndrome is a genetic condition in females that is a result of abnormal chromosomes. Patients with Turner syndrome are typically short, have abnormal physical features, and lack the physical changes normally associated with puberty. In addition, some patients with Turner syndrome have low bone density (osteoporosis) and differences in learning abilities.

This study will research the effects of steroid hormones on patients with Turner syndrome. It will look closely at how taking steroid hormones effects the patient's rate of growth as well as the patient's ability to learn. In addition the study will investigate how different hormones (androgen and estrogen) work when given together as a combination.

All patients asked to participate in this study will receive growth hormone injections. However, half of the patients will receive an additional sex steroid hormone (oxandrolone) in the form of a pill. The other half of the patients will receive a placebo or "sugar pill". This will allow the researchers to determine if the combination of the hormones produces different results than growth hormone alone.

The study will last approximately 2 years. After 2 years of research the patients may qualify for an additional 2 years of treatment. Patients may benefit directly from this research with increased growth and improved ability to learn.

DETAILED DESCRIPTION:
Turner syndrome is associated with short stature, multiple physical stigmata, and absent pubertal development. We propose to: (1) examine the effects of sex steroids (androgen) on multiple variables (growth rate, GH binding protein, IGF-I, and cognitive function), in the setting of supplemental growth hormone administration and (2) to investigate any synergistic or additive effects of the androgen and estrogen combination on the above variables.

ELIGIBILITY:
* INCLUSION CRITERIA:

Girls with Turner syndrome will qualify to participate in this study if they meet the following criteria:

Karyotype diagnosis compatible with Turner syndrome.

No treatment with estrogen, androgen or growth hormone exceeding twelve months, and no treatment with either of these agents in the preceding 3 months.

Chronological age of 10.0 to 14.9 years.

Bone age less than or equal to 12 years.

EXCLUSION CRITERIA:

Prior treatment with estrogen, androgen, or growth hormone for more than twelve months.

Y component in peripheral karyotype.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 1992-12-11; Study Completion 2007-10-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Palmer CG, Reichmann A. Chromosomal and clinical findings in 110 females with Turner syndrome. Hum Genet. 1976 Dec 29;35(1):35-49. doi: 10.1007/BF00295617. PMID 1002163